CLINICAL TRIAL: NCT05466643
Title: A Multicenter, Randomized, Placebo-controlled Clinical Trial to Evaluate the Efficacy and Safety of DWP16001 as add-on Therapy to Drug A, With or Without Antihyperglycemic Drugs, in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study to Investigate the Effect of DWP16001 as add-on Therapy to Drug A in Patients With Type 2 Diabetes Mellitus
Acronym: ENHANCE-I
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DW_DWP16001305
Record Dates: First submitted 2022-07-12; First posted 2022-07-20 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Enavogliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DWP16001 (Experimental)
  Interventions: Drug: DWP16001 0.3mg
- Placebo (Placebo Comparator)
  Interventions: Drug: DWP16001 Placebo

INTERVENTIONS:
Drug: DWP16001 0.3mg — 1 tablet, Orally, Once daily single dose
  Arms: DWP16001
Drug: DWP16001 Placebo — 1 tablet, Orally, Once daily single dose
  Arms: Placebo

SUMMARY:
A multicenter, randomized, placebo-controlled clinical trial, double-blind, parallel-group

DETAILED DESCRIPTION:
Phase 3 study in patients with T2DM, who have inadequate glycemic control on Drug A alone or Drug A in combination with antihyperglycemic drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥19 and ≤ 80 years of age at Visit 1 (Screening) in accordance with American Diabetes Association (ADA) guidelines
2. Patients who had received a stable dose of Drug A for at least 8 weeks prior to Visit 2 (Run-in vis it).
3. In case of antidiabetic concomitant medications, patients who have maintained up to 2 oral antidiabetic drugs [OADs]) without changing regimen/dose/dosage at least 8 weeks prior to Visit 2 (Run-in visit).
4. Patients with FPG of <270 mg/dL at Visit 1 (Screening) (FPG result at Visit 1 will use local laboratory results)
5. Body Mass Index (BMI) 18.0-40.0 kg/m2.

Exclusion Criteria:

1. Patients with type 1 diabetes mellitus (T1DM), congenital diabetes mellitus (DM), or secondary diabetes as follows:

   1. Diabetes caused by Cushing's syndrome and acromegaly.
   2. Patients with fasting C-peptide <0.70 ng/mL (0.23 nmol/L) are excluded if the Investigator cannot rule out T1DM based on the clinical assessment.
   3. Patients with a history of T1DM or a history of ketoacidosis or patients assessed by the Investigator as possibly having T1DM confirmed with a C-peptide <0.70 ng/mL (0.23 nmol/L).
   4. History of other specific types of diabetes (eg, genetic syndromes, secondary pancreatic diabetes, diabetes due to endocrinopathies, drug- or chemical-induced, and post-organ transplant).
2. Patients receiving SGLT2 inhibitors, GLP-analogues, thiazolidinediones, or sulfonylureas (at Screening and Run in).
3. At Visit 1 (Screening), patients with a history of the following:

   1. Patients who had experienced severe hypoglycemia within 24 weeks prior to Screening or who had experienced hypoglycemia at least 3 times a week within 8 weeks prior to Screening.
   2. Patients with a history of diabetic ketoacidosis or coma from hyperosmolar hyperglycemic syndrome within 24 weeks.
   3. Patients with a history of myocardial infarction, unstable angina, arterial revascularization, stroke, transient ischemic attack, within 3 months prior to Screening.
   4. Patients with New York Heart Association (NYHA) Class III, IV congestive heart failure or arrhythmia requiring treatment. History of dose modification of a treatment for thyroid dysfunction within the past 6 weeks (If patients have been on a stable dose from before enrollment to the study, concomitant administration is allowed. Dose reduction for stable condition is allowed).
   5. Patients who had a surgical operation within 4 weeks (excluding minor surgeries without restriction on food and fluid intake) or who are scheduled to have a significant surgery during the study period.
   6. Patients with pituitary insufficiency or adrenal insufficiency.
   7. Patients with pulmonary embolism, severe pulmonary dysfunction, or who are susceptible to be accompanied by hypoxemia at Screening.
4. Patients who are on or likely to require treatment for ≥14 consecutive days or repeated courses of pharmacologic doses of corticosteroids.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes from Baseline HbA1c | at Week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hong JH, Min KW, Lee CB, Chamnan P, Sirirak T, Sony K, Sattanon S, Kim HJ, Kim SY, Kim Y, Heo JA, Cho JM, Nah JJ, Park MH, Kim JH. Efficacy and Safety of Enavogliflozin as Add-on in Adults with Type 2 Diabetes Mellitus Inadequately Controlled with Insulin or Insulin with Other Antidiabetic Drugs. Diabetes Metab J. 2025 Dec 15. doi: 10.4093/dmj.2025.0477. Online ahead of print. PMID 41397686